CLINICAL TRIAL: NCT02911467
Title: Magnetic Resonance (MR) Imaging With Hyperpolarized Pyruvate (13C) as a Predictive Biomarker of Response to Androgen Signaling Inhibitors in Castration-Resistant Prostate Cancer
Brief Title: Magnetic Resonance (MR) Imaging With Hyperpolarized Pyruvate (HP) (13C) in Castration-Resistant Prostate Cancer
Acronym: MR
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Low Accrual
Sponsor: Rahul Aggarwal (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Rahul Aggarwal, Rahul Aggarwal, MD, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 15559; 5R01CA166655-04 (NIH)
Record Dates: First submitted 2016-09-19; First posted 2016-09-22 (Estimated); Last update posted 2020-07-24 (Actual); Status verified 2020-07

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Pyruvic Acid; Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- MR imaging with hyperpolarized 13C pyruvate of men with CRPC (Experimental): 75 men with castration-resistant prostate cancer (CRPC) will undergo MR imaging with hyperpolarized 13C pyruvate of a pre-selected target lesion at baseline and after 1 month of treatment with an androgen signaling inhibitor. Patients with CRPC that is not primarily refractory (defined as disease progression by PCWG2 criteria within 6 months of treatment initiation) to Androgen Signaling Inhibitors (ASI) treatment will undergo a third metabolic MR scan at the time of disease progression. Patients may undergo optional MR- or CT-guided tumor biopsies at baseline and at the time of disease progression.
  Interventions: Drug: Pyruvate (13C); Device: MRI

INTERVENTIONS:
Drug: Pyruvate (13C) — Pyruvate injection followed by an MRI scan.
  Other Names: Hyperpolarized Pyruvate (13C)
Device: MRI — MRI scan following the Pyruvate injection
  Other Names: Magnetic Resonance Imaging

SUMMARY:
This is a prospective imaging study evaluating the utility of baseline metabolic MR imaging with Hyperpolarized Pyruvate (HP) (13C) as a predictive response biomarker to androgen signaling inhibition in patients with castration-resistant prostate cancer.

DETAILED DESCRIPTION:
This is a prospective imaging study evaluating the utility of baseline metabolic MR imaging as a predictive response biomarker to androgen signaling inhibition in patients with castration-resistant prostate cancer. Patients with a target lesion that is amenable for metabolic MR imaging will be eligible for study participation. Patients will undergo baseline metabolic MR imaging with Hyperpolarized Pyruvate C-13 pyruvate followed by initiation of androgen signaling inhibition (either as standard of care or as part of clinical trial; including abiraterone and/or enzalutamide treatment). Patient will subsequently undergo repeat metabolic MR scan after 28 days (+/- 7 days) of therapy. For those without primarily refractory disease, a third metabolic MR scan will be completed at the time of radiographic disease progression by The Prostate Cancer Clinical Trials Working Group 2 (PCWG2) criteria. MR- or CT-guided tumor biopsies are optional at baseline and at the time of disease progression.

ELIGIBILITY:
Inclusion Criteria:

1. Biopsy-proven prostate cancer.
2. Progressive, castration-resistant disease according to PCWG2 criteria.
3. Planned treatment with an androgen signaling inhibitor (e.g., abiraterone, enzalutamide, apalutamide (ARN-509)). Patients must not be receiving androgen signaling inhibitor at the time of the baseline MR scan. Combination treatment (e.g., androgen signaling inhibitor in conjunction with another systemic treatment) is allowed.
4. Presence of at least one target lesion detected by standard staging scans that, in the judgment of Study Investigators, would be amenable to hyperpolarized C-13 pyruvate/metabolic MR imaging:

   * Soft tissue/visceral organ target lesions must measure at 1.5 cm in long axis diameter on CT or MRI.
   * Target lesions in the bone must be visualized by CT or MRI (lesions present only on bone scan do not qualify).
   * For patients with target lesion in prostate/prostatic bed:

     i. No contra-indications to endorectal coil insertion (e.g., patients with a prior abdominoperineal resection of the rectum or latex allergy).

   ii. No prior local treatment to the selected lesion. Patients who have received prior radiation or ablative therapy to the prostate will be required to have biopsy-proven evidence of disease recurrence following completion of local therapy.
5. The subject is able and willing to comply with study procedures and provide signed and dated informed consent.
6. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
7. Adequate organ function, including absolute neutrophil count (ANC) ≥ 1500 cells/µL, hemoglobin ≥ 9.0 gm/dL, platelets ≥ 75,000 cells/µL, creatinine < 1.5 x ULN or estimated creatinine clearance ≥ 50 mL/min (by the Cockcroft Gault equation), bilirubin <1.5x ULN (unless Gilbert's is suspected in which case total bilirubin < 3 x ULN), aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 1.5x ULN.
8. For patients undergoing optional tumor biopsy:

   * No history of bleeding diathesis.
   * Patients on anti-coagulation they must be able to safely stop treatment for purposes of tumor biopsy.
9. For patients with partners of childbearing potential, willing to use adequate contraception for one month after undergoing HP pyruvate infusion.
10. Patients must have prior bilateral orchiectomy or be on continuous luteinizing-hormone releasing hormone (LHRH) analogue therapy for the duration of study.
11. Castrate level of serum testosterone (< 50 ng/dL) at study entry.

Exclusion Criteria:

1. Patients who because of age, general medical or psychiatric condition, or physiologic status cannot give valid informed consent.
2. Patients unwilling or unable to undergo MR imaging, including patients with contra-indications to MRI, such as cardiac pacemakers or non-compatible intracranial vascular clips.
3. Metallic hip implant or any other metallic implant or device that distorts local magnetic field and compromises the quality of MR imaging.
4. Poorly controlled hypertension, defined as systolic blood pressure at study entry greater than 160 mm Hg or diastolic blood pressure greater than 100 mm Hg. The addition of anti-hypertensives to control blood pressure is allowed.
5. Congestive heart failure or New York Heart Association (NYHA) status ≥ 2.
6. A history of clinically significant EKG abnormalities, including QT prolongation (QTcF > 500 ms), a family history of prolonged QT interval syndrome, or myocardial infarction (MI) within 6 months of study entry. Patients with rate-controlled atrial fibrillation/flutter will be allowed on study.
7. Any condition that, in the opinion of the Principal Investigator, would impair the patient's ability to comply with study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2016-11-08 (Actual); Primary Completion 2020-07-20 (Actual); Study Completion 2020-07-20 (Actual)

PRIMARY OUTCOMES:
Mean difference in baseline intra-tumoral peak lac/pyr ratio on HP C-13 MRI in ASI-refractory versus ASI-responsive CRPC tumors | Up to 6 months
  ASI-refractory disease is defined as progression by PCWG2 criteria within 6 months of treatment initiation. ASI-responsive disease includes all other tumors not meeting this criterion. A two sample t-test will be used to compare the mean intra-tumoral HP lac/pyr ratio between treatment-refractory versus treatment-responsive tumors. If a non-parametric distribution is observed, a Mann-Whitney test may also be used to compare the two groups.

SECONDARY OUTCOMES:
Association between change from baseline in peak intra-tumoral HP lac/pyr ratio after 28 days of ASI treatment with subsequent clinical outcomes on ASI treatment | Up to 28 days
  For the purposes of analyzing the association between early change in lac/pyr ratio on HP MRI with subsequent clinical outcomes, the cohort will be dichotomized according to whether follow up scan 4 weeks (28 days) after starting treatment demonstrates increase versus decrease in peak intratumoral lac/pyr ratio compared to baseline. The Prostate-specific antigen (PSA) response rate (PCWG2 criteria) will be compared between dichotomized groups using the chi-squared test. The log rank test will be used to compare the radiographic progression-free survival between the two groups
Mean percent change from baseline in peak intra-tumoral HP lac/pyr ratio on repeat metabolic MRI | Up to 6 months
  The mean percent change from baseline in peak intra-tumoral HP lac/pyr ratio to repeat metabolic MRI obtained at the time of radiographic disease progression by PCWG2 criteria will be descriptively reported for the entire study cohort and for the subgroups of patients with treatment- refractory and treatment-responsive prostate cance
Baseline peak intra-tumoral HP lac/pyr ratio cut-point that most accurately predicts for response versus refractoriness to subsequent ASI treatment | Baseline
  Receiver-operating-curve will be applied to determine the optimal cut-point of peak intra-tumoral lac/pyr values on MRI that accurately distinguish treatment-refractory versus treatment responsive prostate cancer.
Frequency of clinically significant changes in safety variables over time | Up to 6 months
  Safety endpoints include monitoring for the occurrence of treatment-emergent AEs. Toxicities will be graded using the National Cancer Institute (NCI) Common Terminology (Toxicity) Criteria for Adverse Events (CTCAE) version 4.0
Mean Intra-patient reproducibility of HP lac/pyr ratio | Up to 6 months
  Intra-patient reproducibility of HP lac/pyr ratio for patients who undergo repeated dose imaging studies, as descriptively reported using summary statistics

CONTACTS AND LOCATIONS:
Overall Officials: Rahul Aggarwal, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2019-07-10): https://cdn.clinicaltrials.gov/large-docs/67/NCT02911467/ICF_000.pdf